CLINICAL TRIAL: NCT05414292
Title: Impacts of Mechanistic Target of Rapamycin (mTOR) Inhibition on Aged Human Muscle.
Brief Title: Impacts of Mechanistic Target of Rapamycin (mTOR) Inhibition on Aged Human Muscle (Rapamune)
Acronym: Rapamune
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Philip Atherton, Professor, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Rapamune_COMAP
Record Dates: First submitted 2022-05-30; First posted 2022-06-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Muscle Atrophy; Age-Related Sarcopenia
MeSH Terms: conditions — Muscular Atrophy | interventions — Sirolimus; Tablets; Resistance Training

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will not know if they are taking Rapamune or placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug group (Experimental): Will take 1mg Rapamune (sirolimus) in oral tablet form daily for 16 weeks.
  Interventions: Drug: Rapamune (sirolimus) 1Mg Tablet; Behavioral: Unilateral resistance exercise training
- Placebo group (Placebo Comparator): Will take a placebo tablet (lactose) daily for 16 weeks
  Interventions: Behavioral: Unilateral resistance exercise training

INTERVENTIONS:
Drug: Rapamune (sirolimus) 1Mg Tablet — Take Rapamune to see the effect on muscle structure and function during a 14 week unilateral resistance exercise training programme.
  Other Names: Rapamycin; Sirolimus; Rapamune
  Arms: Drug group
Behavioral: Unilateral resistance exercise training — Participants will complete unilateral leg extension resistance training 3 times per week for 14 weeks at 75% of their 1 repetition maximum
  Other Names: Leg extension; Strength training

SUMMARY:
As people age, muscle mass and function is lost and exercise training is an important way to reduce the effects of this and remain independent. However, not everyone can perform this exercise and the muscle responses to exercise are often reduced in older people. So far there has been no drug found to specifically treat or reduce this problem.

Muscle size depends on the balance of muscle protein breakdown and synthesis (building). This balance is regulated by multiple signals within the body, but a particular molecule - the mechanistic target of rapamycin (mTOR), is known to play an important role. For protein synthesis to build up the muscles, this pathway is needed to start the process when triggered by eating protein or exercise. Although this would suggest that mTOR activity is good, excessive levels of this signalling seem to have negative impacts on muscle maintenance with age.

In animal studies, blocking mTOR signalling has stopped the development of a number of age-related diseases and increased health-span. Drugs that block this pathway (e.g. Rapamune) reduce the stimulation of muscle protein synthesis, possibly through changing the immune system, but conversely have also been shown to increase muscle size and reduce markers of nerve supply loss. This means that drugs which block the mTOR pathway could, in older people, help to reduce the negative impacts of excessive mTOR signalling on muscle size and function.

The investigators aim to recruit 16 healthy male volunteers over 50 years old to investigate how the drug Rapamune (which blocks the mTOR pathway) affects aged human muscle both on its own and when combined with resistance exercise training.

DETAILED DESCRIPTION:
Skeletal muscle is known for its role in locomotion however, muscles are also important for maintaining whole-body metabolic health. Skeletal muscles represent a vast protein store, the amino acids from which can be broken down in times of fasting, infection and disease in order to provide energy and amino acids to maintain other critical organs. With increases in the ageing population, this will inevitably increase age-related co-morbidities, and also the prevalence of frailty and increased healthcare costs.

A major facet of frailty is skeletal muscle atrophy and loss of function, and critically, these are associated with poorer clinical outcomes (e.g. surgery), so mitigating age-related muscle loss is crucial for healthy ageing. The processes of muscle loss with ageing in humans are a combination of neurodegeneration of lower motor neurons and concomitant muscle fibre atrophy. While the underlying mechanisms of age-related muscle loss are unclear, a reduced responsiveness to key environmental cues, namely nutrition and movement ("anabolic resistance"), would appear to be central. To date, no pharmaceuticals have yielded the necessary safety and efficacy effects to mitigate age-related muscle loss so exercise, particularly resistance exercise training (RET), remains the most established intervention to improve muscle mass and function in older people. Nonetheless, not all older people can perform RET, and muscle growth responses to RET are diminished in older age. As such, the search for interventions to mitigate muscle ageing and maximise responses to exercise pre-/rehabilitation in terms of muscle growth and function remain key.

The mechanistic target of rapamycin (mTOR) is often termed a "master regulator" in relation to skeletal muscle homeostasis and exists in two distinct complexes, mTORc1 and mTORc2. The most established role of mTORc1 in muscle is as a cellular sensor of nutrients and movement, where signals are conveyed to mTOR substrates, regulating the rate of mRNA translation and thus muscle protein synthesis (MPS). mTOR activity is required for the stimulation of MPS by intake of dietary proteins or free amino acids, in addition to contractile activity, and as such is commonly thought of as being positive in relation to muscle mass. Additionally, administration of rapamycin (a naturally occurring compound that inhibits mTORc1) alongside exercise or nutrient-intake has been shown to reduce the stimulation of MPS. However, confounding the notion of a positive role of mTOR on skeletal muscle, hyper-activation of mTOR has been shown in both ageing rodent and human muscle, suggesting that mTOR signalling has negative impacts in relation to muscle maintenance in ageing.

Despite the positive effects of mTOR in relation to the stimulation of MPS, in animal models data suggest that pharmacological attenuation of mTOR signalling can counteract several age-related diseases and co-morbidities, and increase overall health-span. The major negative ageing traits found to be lessened by dampening mTOR signalling (i.e. with rapamycin) are related to the immune system, organ morphology, neo-plastic disease and neurological dysfunction e.g. motor control. From these studies, the beneficial effects of rapamycin on health-span are clear, but this contrasts the positive impacts mTOR signalling have on muscle. Inhibition of mTOR would be predicted to negatively impact muscle protein turnover however, this is not the case.

Indeed, recent work has challenged the notion of mTOR suppression negatively impacting skeletal muscle metabolism in a number of experimental settings. In pre-clinical models of ageing and/or muscle dysfunction, long-term administration of rapamycin did not negatively impact skeletal muscle mass in mice treated with rapamycin across the life-course. Additionally, long-term administration of rapamycin (9-22 months), showed a mitigation of muscle mitochondrial ageing, reflected by markers of mitochondrial DNA genome stability. Perhaps the most compelling evidence of rapamycin benefiting ageing muscle is from a study where rapalog (a rapamycin analog) treatment was administered to mice where hyper-active mTOR signalling was observed in aged sarcopenic animals, as is also shown in older humans. Crucially, following Rapalog treatment animals demonstrated increases in muscle fibre area in addition to a down-regulation of cellular senescence markers and genes associated with neuromuscular denervation. These works challenge the notion that in older age with mTOR hyper-activation, mTOR-inhibition would have negative effects, and it is now accepted that ageing and age-associated diseases that arise from hyperactive mTORC1 signalling may benefit from mTOR inhibitors. As such, insight into the effects of mTORc1 inhibition are needed in humans, especially in the context of "anabolic resistance", which limits both muscle maintenance and growth potential in older adults. As an immunosuppressant, rapamycin may also present benefits for the treatment of COVID-19 which is a current highly important area of emerging research.

In this study the participant will have muscle size, function and metabolism measured over a 16 week period while either taking the drug Rapamune or a placebo. They will also complete 14 weeks of unilateral resistance exercise with visits described below.

1. Pre-study Assessment

   Twenty-four hours before attending their main pre-study assessment, participants will be asked to consume the labelled creatine (D3-labelled; Cre) and (D3) methylhistidine (3-MH) tracers.. In order to trace these tracers into urine and plasma body pools respectively, participants will be asked to provide a urine sample before consuming these tracers (which they will bring with them the following day), and the blood sample from screening will be used for 3-MH analysis to minimise participant burden. In the 24-hours between consuming the tracer drink and attending for their pre-study assessment participants will be asked to collect all urinary output for which containers will be provided. Participants will also be asked to collect spot urine samples at ~48 amd 72-hours after consuming the tracer drink.

   For their main pre-study assessment, participants will be randomly assigned to either a rapamycin inhibitor (Rapamune) or placebo (matching benign capsule containing sugar to achieve as equal weight and appearance to the treatment product as possible) group (single-blind), and will report to the laboratory for their pre-study assessment day. A suite of baseline assessments will then be performed including body composition (e.g. MRI and muscle ultrasound to determine lean mass, fat mass, muscle thickness, cross-sectional area (CSA) and muscle architecture) and measures of muscle strength and function (1-RM, MVC, power, SPPBT and iEMG). These measures will be repeated throughout the intervention period to monitor temporal changes. Throughout this visit, 6 venous blood samples (~5 ml) will be taken for the assessment of muscle protein breakdown (MPB) via the 3-MH tracer consumed the previous day.

   At the end of their pre-study assessment visit, participants will begin a two week lead-in phase of Rapamune or placebo capsules. On day 13-15 of this lead-in phase, participants will attend the laboratory for their muscle biopsies (~150 mg each), which will be collected from the vastus lateralis (VL) of both legs (rest and exercise). This bilateral biopsy collection will allow volunteers to act as their own controls by providing both an exercise trained leg and a rested leg; to also compare the effects of Rapamune combined with contractile stimulus. Biopsy sites will be closed by sutures, which are removed (and the wound site checked) after 5-7 days. After these initial biopsies, participants will be given their bolus dose of D2O to begin assessing rates of MPS. To minimise the risk of dizziness from D2O consumption, this initial dose will be split into 6-8 smaller does provided throughout the day. Two hours after their final D2O dose, participants will be asked to provide a saliva sample..
2. Resistance exercise training (RET) RET consisting of unilateral knee-extension exercise (i.e. 6 × 8 repetitions at 75% of one repetition maximum (1-RM)) will be performed 3 x each week 14-weeks.The RET will be progressive, with reassessment of 1-RM being performed at regular intervals to maintain exercise intensity. Participants will also be provided with their interventional drug (for daily dosing) and D2O tracer top-ups (for the assessment of MPS) on a weekly basis during these visits, with a venous blood sample also collected weekly. Participants will be asked to collect daily saliva samples for the first week (~2h after D2O consumption), and on a weekly basis thereafter.
3. Mid-study Assessment 1 After 3-weeks of RET, all of the baseline procedures from the pre-study assessment visits will be repeated, with the exception of the measures relating to the D3 and 3-MH tracers, and MRI which will not be performed on this visit.
4. Mid-study Assessment 2 After 6-weeks of RET, all of the baseline procedures from the pre-study assessment visits will be repeated. No further D2O will be given or saliva samples collected after week 6 of RET.
5. Post-study Assessment After 14-weeks of RET, all of the baseline procedures from the pre-study assessment visits will be repeated. The label of the creatine will be 13C instead of D3 to permit a second analysis of whole body muscle mass.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Participant is physically able to complete the resistance exercise training programme

Exclusion Criteria:

* • A BMI <18 or >35 kg/m2

  * Active cardiovascular, cerebrovascular or respiratory disease: e.g. uncontrolled hypertension (BP > 160/100), angina, heart failure (class III/IV), arrhythmia, right to left cardiac shunt, recent cardiac event, COPD, pulmonary hypertension or recent stroke
  * Any metabolic disease
  * Clotting dysfunction
  * A history of, or current neurological or musculoskeletal conditions (e.g. epilepsy)
  * Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance (this must remain for ALL UoN FMHS UREC approved studies)
  * Contraindications to MRI scanning including claustrophobia, pacemaker, metal implants etc. which will be assessed through an MRI safety screening questionnaire.
  * Contraindications to the use of Rapamycin e.g. those due scheduled vaccinations (as rapamycin can reduce the efficacy of vaccines).

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in muscle mass from baseline | 0 and 16 weeks
  To determine the impacts of rapamycin, an mTOR inhibitor, on human muscle mass through whole body muscle mass measures by MRI and D3 creatine tracer, and ultrasound of the thigh muscles.
Change in muscle mass from baseline | 0 and 8 weeks
  To determine the impacts of rapamycin, an mTOR inhibitor, on human muscle mass through whole body muscle mass measures by MRI and D3 creatine tracer, and ultrasound of the thigh muscles.
Change in muscle mass from baseline | 0 and 5 weeks
  To determine the impacts of rapamycin, an mTOR inhibitor, on human muscle mass through whole body muscle mass measures by MRI and D3 creatine tracer, and ultrasound of the thigh muscles.

SECONDARY OUTCOMES:
Change in muscle strength | 0, 5, 8 and 16 weeks
  To determine the impacts of rapamycin on muscle function through muscle strength measures of 1 Repetition Maximum
Change in muscle power | 0, 5, 8 and 16 weeks
  To determine the impacts of rapamycin on muscle function through muscle power measured from countermovement jump analysis.
Change in muscle function | 0, 5, 8 and 16 weeks
  To determine the impacts of rapamycin on muscle function through muscle performance measures included in the short performance physical battery test (SPPBT).
Change in neuromuscular function | 0, 5, 8 and 16 weeks
  • To determine the impacts of rapamycin on muscle function through muscle-nerve electrical signals studied with electromyography (EMG).
Change in Muscle Protein Synthesis | 2, 5, and 8 weeks
  To determine the impacts of rapamycin on muscle metabolism through effects on muscle protein synthesis (via D2O tracer) from muscle biopsies.
Change in Muscle Protein Breakdown | 2 and 16 weeks
  To determine the impacts of rapamycin on muscle metabolism through effects on muscle protein breakdown (via 3-MH tracer) obtained from muscle biopsies.
Immune function | 0, 2, 5, 8 and 16 weeks
  Collection of peripheral blood mononuclear cells to study the immune cytokine profile using an Isoplexis system

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham School of Medicine, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data may be shared with collaborators including anthropometric data and samples where consent is given for this.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The data will be available on conclusion of the study.
Access Criteria: Listed collaborators will have access on request with data given on approval by the principal investigator